CLINICAL TRIAL: NCT01347333
Title: Phase IV Trial Evaluating the Use of Stereotactic Body Radiotherapy for the Treatment of Liver Metastases and Primary Liver Tumors
Brief Title: Stereotactic Body Radiotherapy for Liver Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Kathy Baglan, MD, Radiation Oncologist, Mercy Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-045
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Liver Metastases; Hepatocellular Carcinoma; Intrahepatic Cholangiocarcinoma
Keywords: liver metastases; stereotactic radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- liver metastases (Other): Oligometastases (1-3) with aggregate tumor diameter < 6 cm Metastases from neuroendocrine tumors with functional endocrine syndromes
  Interventions: Radiation: Stereotactic body radiosurgery
- Primary Liver Tumors (Other): Hepatocellular Carcinoma Intrahepatic Cholangiocarcinoma
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiosurgery — 36-60 Gy / 3 fractions (12-20 Gy per fraction) OR 45-50 Gy / 5 fractions (9-10 Gy per fraction)
  Arms: liver metastases
Radiation: Stereotactic Body Radiotherapy — 26-30 Gy / 1 fraction OR 36-45 Gy / 3 fractions (12-15 Gy per fraction) OR 40-50 Gy / 5 fractions (8-10 Gy per fraction)
  Arms: Primary Liver Tumors

SUMMARY:
This study will evaluate the local control rate as well as acute and late toxicity rates of stereotactic body radiotherapy for the treatment of liver metastases and unresectable primary liver tumors such as hepatocellular carcinoma and intrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
This study is a single site, non-randomized, prospective, phase IV trial.

Composed of 4 patient groups:

1. Oligometastases (1-3) with aggregate tumor diameter < 6 cm
2. Metastases from neuroendocrine tumors with functional endocrine syndromes
3. Unresectable hepatocellular carcinoma (HCC)
4. Unresectable intrahepatic cholangiocarcinoma (IHCC) Data collected will include patient demographics, pathology data, tumor stage, SBRT dose fractionation scheme, dose received by adjacent critical normal tissues, tumor recurrence data, and acute and late toxicities. Follow up data will be collected during the patient's standard office visits. The anticipated duration of this study is 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >= 18 years
* Zubrod performance status of 0-3
* Oligometastases (1-3) with aggregate tumor diameter < 6 cm
* Metastases from neuroendocrine tumors with functional endocrine syndromes for symptom palliation
* Unresectable hepatocellular carcinoma (HCC)
* Unresectable intrahepatic cholangiocarcinoma (IHCC)
* Maximum tumor diameter < 6 cm
* Adequate liver function:

Total bilirubin < 3 mg/dL Serum albumin > 2.5 g/dL Serum levels of liver enzymes < 3 times the upper limit of normal Normal PT and PTT unless patient is receiving anticoagulant medication

- Signed study-specific consent form

Exclusion Criteria:

* Maximum tumor diameter > 6 cm
* Prior radiotherapy to the liver
* Pregnant or lactating women, due to potential exposure of the fetus to RT and unknown effects of RT on lactating females
* Patients with psychiatric or addictive disorder that would preclude obtaining informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany G Sleckman, MD, Study Director — Mercy Hospital St. Louis
Locations (1):
- St. John's Mercy Medical Center, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liver Metastases | Primary Liver Tumors
Started | 23 | 0 (No participants were enrolled in the Primary Liver Tumor arm.)
Completed | 23 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were analyzed in primary liver tumors because none were enrolled to that group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liver Metastases | Primary Liver Tumors | Total
Number analyzed (Participants) | 23 | 0 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 15 |  | 15
  >=65 years | 8 |  | 8
Age, Continuous [Median (Full Range); unit: years] | 63 [47 to 79] |  | 63 [47 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 |  | 12
  Male | 11 |  | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 0 | 23

OUTCOME MEASURES:

1. Primary Outcome: Local Tumor Recurrence Rate
Description: Primary endpoint will be local tumor recurrence rate. Local recurrence is defined as tumor recurrence within the planning target volume.
Time Frame: 5 years
Population: No patients enrolled into primary liver tumor group.
Measure: Count of Participants; unit: Participants
Arm/Group | Liver Metastases | Primary Liver Tumors
Number analyzed (Participants) | 23 | 0
Participants | 4 | 0

2. Secondary Outcome: Late Complication Rates
Description: Toxicities will be assessed using CTCAE grading criteria at specified timepoints.
Time Frame: 5 years
Population: This outcome was not collected.
Arm/Group | Liver Metastases | Primary Liver Tumors
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Description: At risk for primary liver tumor is 0 because no patients were enrolled to this group.
Arm/Group | Liver Metastases | Primary Liver Tumors
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/0
Other Adverse Events (participants affected / at risk) | 0/23 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No